CLINICAL TRIAL: NCT00834119
Title: Assessment of the Effectiveness of Regular Use of Intranasal Steroids in Alleviating Nasal Symptoms in Allergic Rhinitis When Used Alone or in Combination With Oral Antihistamine
Brief Title: Assessment of Intranasal Steroids in Allergic Rhinitis When Used Alone or in Combination With an Oral Antihistamine (Study P03270)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03270
Record Dates: First submitted 2008-10-30; First posted 2009-02-03 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone furoate (Experimental)
  Interventions: Drug: Mometasone furoate
- Mometasone furoate plus an oral antihistamine (Experimental)
  Interventions: Drug: Mometasone furoate

INTERVENTIONS:
Drug: Mometasone furoate — Mometasone furoate 200 mcg (2 puffs in each nostril) once a day for 28 days
  Other Names: Nasonex; SCH 32088
  Arms: Mometasone furoate
Drug: Mometasone furoate — Mometasone furoate 200 mcg (2 puffs in each nostril) once a day plus an oral antihistamine added at Day 28 (Visit 2) at the discretion of the physician
  Other Names: Nasonex; SCH 32088
  Arms: Mometasone furoate plus an oral antihistamine

SUMMARY:
This is a Phase 4, non-comparative, open-label, multi-center study. It is designed to determine the effectiveness of regular intranasal steroid use in alleviating allergic rhinitis nasal symptoms, when used alone or in combination with an oral antihistamine. Subjects will receive 200 mcg (2 puffs in each nostril) of mometasone furoate once a day. An oral antihistamine at the discretion of the physician may be added at Day 28 (Visit 2), if patients fail to improve nasal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent form
* Subjects must be between 18-65 years of age, of either sex and any race
* Subjects must be diagnosed by the physician to have moderate to severe allergic rhinitis according to ARIA guidelines.
* Subjects must be mometasone furoate naïve.

Exclusion Criteria:

* Significant comorbid medical condition.
* Respiratory tract infection.
* Any contraindications according to mometasone furoate product monograph.
* Patients who have received antihistamine treatment within the last 5 days.
* Patients who have received corticosteroid treatment within the last 30 days.
* Patients who are likely to require the administration of systemic steroids during the course of this program.
* Any condition which in the doctor's opinion could interfere with the patient completion of this program.
* Pregnant or lactating patients.
* Patients with local infections involving the nasal mucosa.
* Patients with structural abnormalities or who have undergone nasal surgery or trauma in the past 6 months.
* Patients with hypersensitivity to mometasone furoate or are allergic to corticosteroids.
* Patients who are prone to nose bleeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-09-01 (Actual); Primary Completion 2004-04-01 (Actual); Study Completion 2004-04-01 (Actual)

PRIMARY OUTCOMES:
To assess the mean change in total nasal symptom score from Baseline to the Final Visit of regular intranasal steroid use (mometasone furoate) in allergic rhinitis patients when used alone or in combination with an oral antihistamine. | Day 28 and Day 56

SECONDARY OUTCOMES:
Patient satisfaction with intranasal steroid monotherapy. | Day 28
Potential benefit of an oral antihistamine in combination with an intranasal steroid | Day 56